CLINICAL TRIAL: NCT02969915
Title: Strategies to Improve the HIV Care Continuum Among Key Populations in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); YR Gaitonde Centre for AIDS Research and Education (Other); Elton John AIDS Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00082575; R01DA041034 (NIH); K24DA035684 (NIH)
Record Dates: First submitted 2016-11-18; First posted 2016-11-21 (Estimated); Results first posted 2022-12-22 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
Keywords: people who inject drugs; men who have sex with men; HIV; India
MeSH Terms: conditions — HIV Infections; Homosexuality | interventions — Fertility

STUDY DESIGN:
Intervention Model Description: Matched-pair cluster-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated care centers (Active Comparator): Participants in the active comparator arm have access to integrated care centers (ICCs)
  Interventions: Behavioral: Integrated Care Centers
- ICC + incentives (Experimental): Participants in the experimental arm have access to the ICC intervention and the incentive intervention
  Interventions: Behavioral: Incentives; Behavioral: Integrated Care Centers

INTERVENTIONS:
Behavioral: Incentives — Treatment incentives are offered to HIV-positive participants for reaching treatment targets, including retention to medical follow-up, initiating antiretroviral therapy, and maintaining high adherence with antiretroviral therapy.
  Other Names: ICC+
  Arms: ICC + incentives
Behavioral: Integrated Care Centers — ICCs offer key-population-oriented, vertically-integrated harm reduction, HIV testing, and HIV treatment services
  Other Names: ICC

SUMMARY:
This clinical trial will compare the effectiveness of integrated care centers vs. integrated care centers plus HIV patient treatment incentives for achieving HIV treatment targets among people who inject drugs and men who have sex with men in India. The investigators will also assess cost-effectiveness and barriers and facilitators to implementation through targeted mixed-methods approaches. This study is a model for improving HIV treatment outcomes in key populations in low to middle-income countries.

DETAILED DESCRIPTION:
The trajectory of the HIV epidemic in coming decades will be determined by the degree to which we can identify infected persons and engage them in care - a point implicit in the ambitious UNAIDS "90-90-90" target, which sets 90% goals for HIV diagnosis, linkage of infected persons to sustained antiretroviral therapy (ART), and viral suppression in those treated. Meeting this target requires successful engagement of difficult to reach populations, such as people who inject drugs (PWID) and men who have sex with men (MSM), who bear a disproportionate share of the epidemic, particularly in low to middle income countries. Our team is nearing completion of a multi-site cluster-randomized trial in India to assess the effectiveness of integrated care centers (ICCs) for PWID and MSM compared to usual care. ICC process measures from the first year show robust uptake of HIV counseling and testing, the primary outcome for that trial, but slower than anticipated ART uptake. Demand-side interventions in public health (such as treatment incentives) can be particularly effective when paired with optimized treatment accessibility (i.e., supply). Consequently, the investigators propose to examine whether provision of HIV care and treatment incentives to ICC clients will improve overall utilization of the clinics and downstream HIV care continuum outcomes.

The investigators propose a hybrid effectiveness-implementation design. This will include a 16-site, pair-matched cluster randomized trial to compare the effectiveness of adding of HIV care incentives to ICCs (ICC+) versus standard ICCs on HIV care continuum outcomes, including ART initiation, adherence and viral suppression. Effectiveness will be compared at the ICC level (from a cohort of HIV-infected ART-eligible clients followed in each ICC and process measures deriving from all ICC clients) and at the community-level through a cross-sectional sample accrued via respondent-driven sampling (RDS) 2 years after initiation of the intervention. Because PWID and MSM will be sampled independently from the ICCs in the RDS, it provides an opportunity to characterize outcomes like community viral load and HIV incidence, reflecting impact within the broader PWID/MSM communities. As an exploratory sub-aim, we will use a rigorous scientific design to assess the effects of withdrawing (vs. continuing) incentives beyond the initial intervention phase. Additionally, the investigators will determine the cost-effectiveness of the ICC+ intervention.

ELIGIBILITY:
Inclusion Criteria:

* Speaks Hindi, English, or local language
* HIV-positive
* Antiretroviral therapy (ART) naive or has used ART less than 12 months
* Registered client at the local integrated care center (ICC), which serves either people who inject drugs (PWID) or men who have sex with men (MSM).

Exclusion Criteria:

* Not competent to provide informed consent or participate in the study.
* Receives HIV care in the private sector
* Plans to migrate in next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2314 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shruti H Mehta, PhD, Principal Investigator — Johns Hopkins University; Gregory M Lucas, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- YR Gaitonde Center for AIDS Research and Education, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Yes
The investigators will require prospective collaborators to submit concept sheets to the study PIs that include a brief summary of the proposed hypothesis, summary of research methods, specific data or specimens that are being requested, and plans for analysis. Reasonable requests that address relevant scientific questions will be welcomed and supported to the extent possible.

REFERENCES:
- [Result] Solomon SS, McFall AM, Srikrishnan AK, Verma V, Anand S, Khan RT, Kushwaha BS, Vasudevan C, Saravanan S, Paneerselvam N, Kumar MS, Das C, Celentano DD, Mehta SH, Lucas GM. Voucher incentives to improve viral suppression among HIV-positive people who inject drugs and men who have sex with men in India: a cluster randomised trial. Lancet HIV. 2024 May;11(5):e309-e320. doi: 10.1016/S2352-3018(24)00005-5. Epub 2024 Apr 4. PMID 38583461

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 22 sites were considered for the trial and 16 were selected on the basis of high HIV prevalence. The 16 study sites were matched into pairs and randomized to incentives or usual care. Sites were matched according to key population (people who inject drugs or men who have sex with men) and HIV burden.
Units Other Than Participants: Sites
Groups:
- Incentives: Participants in the experimental arm have access to the ICC intervention and the incentive intervention
  Incentives: Treatment incentives are offered to HIV-positive participants for reaching treatment targets, including retention to medical follow-up, initiating antiretroviral therapy, and maintaining high adherence with antiretroviral therapy.
  Integrated Care Centers: ICCs offer key-population-oriented, vertically-integrated harm reduction, HIV testing, and HIV treatment services
- Usual Care: Participants in the active comparator arm have access to integrated care centers (ICCs)
  Integrated Care Centers: ICCs offer key-population-oriented, vertically-integrated harm reduction, HIV testing, and HIV treatment services
Period: Overall Study
Arm/Group | Incentives | Usual Care
Started | 1114; 8 Sites | 1200; 8 Sites
6-month Follow-up | 901; 8 Sites | 968; 8 Sites
12-month Follow-up | 826; 8 Sites | 885; 8 Sites
18-month Follow-up | 778; 8 Sites | 824; 8 Sites
Completed (24-month follow-up) | 421; 8 Sites | 492; 8 Sites
Not Completed | 693; 0 Sites | 708; 0 Sites
Not completed — Death | 104 | 125
Not completed — Lost to Follow-up | 108 | 112
Not completed — Censored due to COVID-19 | 481 | 471

BASELINE CHARACTERISTICS:
Population: Data are stratified by key population (PWID and MSM). 600 PWID and 514 MSM were at sites assigned to the incentive intervention (1114 total), and 600 PWID and 600 MSM were at sites assigned to usual care (1200 total).
Groups:
- PWID [Usual Care]: People who inject drugs (PWID) in 4 sites assigned to usual care
- PWID [Incentives]: People who inject drugs (PWID) in 4 sites assigned to the incentives intervention
- MSM [Usual Care]: Men who have sex with men (MSM) in 4 sites assigned to usual care
- MSM [Incentives]: Men who have sex with men (MSM) in 4 sites assigned to the incentives intervention
- Total: Total of all reporting groups
Arm/Group | PWID [Usual Care] | PWID [Incentives] | MSM [Usual Care] | MSM [Incentives] | Total
Number analyzed (Participants) | 600 | 600 | 600 | 514 | 2314
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 28 [24 to 33] | 30 [25 to 35] | 30 [25 to 40] | 32 [26 to 40] | 30 [25 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 152 | 0 | 0 | 154
  Male | 598 | 448 | 600 | 514 | 2160
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 600 | 600 | 600 | 514 | 2314
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
HIV RNA <150 copies/mL [Count of Participants; unit: Participants] | 61 | 153 | 108 | 138 | 460
CD4 cell count [Median (Inter-Quartile Range); unit: cells/microliter] — Normal is >/= 500 cells/microliter.
  cells/microliter | 391 [282 to 499] | 384 [242 to 514] | 314 [183 to 477] | 276 [147 to 434] | 347 [210 to 491]
Secondary school education or beyond [Count of Participants; unit: Participants] | 336 | 381 | 375 | 352 | 1444

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Surviving With Viral Suppression
Description: Viral Suppression defined as HIV RNA <150 copies/mL
Time Frame: 12 months
Measure: Number; unit: proportion of participants
Units Other Than Participants: sites
Arm/Group | Incentives | Usual Care
Number analyzed (Participants) | 1114 | 1200
Number analyzed (sites) | 8 | 8
proportion of participants | 0.494 | 0.353
Statistical Analysis 1: Comparison: Incentives vs Usual Care; Test type: Superiority; Risk Ratio (RR) = 1.21, 95% CI 2-sided [0.64 to 2.26]

2. Secondary Outcome: Proportion of Participants Surviving With Viral Suppression
Description: Viral suppression defined as HIV RNA <150 copies/mL
Time Frame: 6 months
Measure: Number; unit: Proportion of participants
Units Other Than Participants: Study sites
Arm/Group | Incentives | Usual Care
Number analyzed (Participants) | 1114 | 1200
Number analyzed (Study sites) | 8 | 8
Proportion of participants | 0.509 | 0.365
Statistical Analysis 1: Comparison: Incentives vs Usual Care; Test type: Superiority; Risk Ratio (RR) = 1.31, 95% CI 2-sided [0.91 to 1.90]

3. Secondary Outcome: Proportion of Participants Surviving With Viral Suppression
Description: Viral suppression defined as HIV RNA <150 copies/mL
Time Frame: 18 months
Population: Overall number of participants analyzed is equal to enrolled cohort minus participants who were censored at the 18-month visit due to COVID-related stoppage.
Measure: Number; unit: Proportion of participants
Units Other Than Participants: Study sites
Arm/Group | Incentives | Usual Care
Number analyzed (Participants) | 1105 | 1166
Number analyzed (Study sites) | 8 | 8
Proportion of participants | 0.497 | 0.358
Statistical Analysis 1: Comparison: Incentives vs Usual Care; Test type: Superiority; Risk Ratio (RR) = 1.16, 95% CI 2-sided [0.70 to 1.95]

4. Secondary Outcome: Proportion of Participants Surviving With Viral Suppression
Description: Viral suppression defined as HIV RNA <150 copies/mL
Time Frame: 24 months
Population: Overall number of participants analyzed is equal to enrolled cohort minus participants who were censored at the 24-month visit due to COVID-related stoppage.
Measure: Number; unit: Proportion of participants
Units Other Than Participants: Study sites
Arm/Group | Incentives | Usual Care
Number analyzed (Participants) | 633 | 729
Number analyzed (Study sites) | 8 | 8
Proportion of participants | 0.471 | 0.325
Statistical Analysis 1: Comparison: Incentives vs Usual Care; Test type: Superiority; Risk Ratio (RR) = 1.29, 95% CI 2-sided [0.85 to 1.95]

5. Secondary Outcome: Proportion of Participants With Viral Suppression at One or More Follow-up Visits
Description: Proportion with viral suppression (HIV RNA <150 copies/mL) at one or more follow-up visits
Time Frame: 24 months
Measure: Number; unit: Proportion of participants
Units Other Than Participants: Study sites
Arm/Group | Incentives | Usual Care
Number analyzed (Participants) | 1114 | 1200
Number analyzed (Study sites) | 8 | 8
Proportion of participants | 0.640 | 0.498
Statistical Analysis 1: Comparison: Incentives vs Usual Care; Test type: Superiority; Risk Ratio (RR) = 1.17, 95% CI 2-sided [0.79 to 1.75]

6. Secondary Outcome: Antiretroviral Therapy (ART) Initiation
Description: Rate of ART initiation among those naive to ART at baseline. This is reported as the proportion of participants who initiated ART.
Time Frame: 12 months
Population: This analysis includes only participants who had never started ART previously
Measure: Number; unit: Proportion of participants
Units Other Than Participants: Study site
Arm/Group | Incentives | Usual Care
Number analyzed (Participants) | 716 | 935
Number analyzed (Study site) | 8 | 8
Proportion of participants | 0.721 | 0.708
Statistical Analysis 1: Comparison: Incentives vs Usual Care; Test type: Superiority; Risk Ratio (RR) = 1.48, 95% CI 2-sided [0.38 to 5.76]

7. Secondary Outcome: Retention to HIV Care
Description: Proportion of participants who attended one or more visits to a government ART clinic in both the 0 to 6 month period and the 6 to 12 month period.
Time Frame: 12 months
Measure: Number; unit: Proportion of participants
Units Other Than Participants: Study site
Arm/Group | Incentives | Usual Care
Number analyzed (Participants) | 1114 | 1200
Number analyzed (Study site) | 8 | 8
Proportion of participants | 0.702 | 0.664
Statistical Analysis 1: Comparison: Incentives vs Usual Care; Test type: Superiority; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.68 to 1.36]

8. Secondary Outcome: ART Adherence
Description: Proportion of participants who had a medication possession ratio of 0.9 or higher after starting ART
Time Frame: 12 months
Measure: Number; unit: proportion of participants
Units Other Than Participants: Study sites
Arm/Group | Incentives | Usual Care
Number analyzed (Participants) | 1114 | 1200
Number analyzed (Study sites) | 8 | 8
proportion of participants | 0.645 | 0.463
Statistical Analysis 1: Comparison: Incentives vs Usual Care; Test type: Superiority; Risk Ratio, log = 1.38, 95% CI 2-sided [0.77 to 2.46]

9. Secondary Outcome: Mortality
Description: All-cause mortality
Time Frame: 12 months
Measure: Number; unit: Proportion of participants
Units Other Than Participants: Study sites
Arm/Group | Incentives | Usual Care
Number analyzed (Participants) | 1114 | 1200
Number analyzed (Study sites) | 8 | 8
Proportion of participants | 0.051 | 0.068
Statistical Analysis 1: Comparison: Incentives vs Usual Care; Test type: Superiority; Risk Ratio (RR) = 0.39, 95% CI 2-sided [0.09 to 1.80]

ADVERSE EVENTS:
Time Frame: 24 months
Description: The research procedures are minimal risk (involve only a blood draw) and the intervention is behavioral. Given these considerations, our reporting obligations for the trial focus only on events that are more likely than not to be associated with i) study procedures, or ii) participation in the intervention. Adverse events are reported through complete (24-month) follow-up.
Arm/Group | Incentives | Usual Care
All-Cause Mortality (participants affected / at risk) | 104/1114 | 125/1200
Serious Adverse Events (participants affected / at risk) | 104/1114 | 125/1200
Other Adverse Events (participants affected / at risk) | 0/1114 | 0/1200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Incentives (N=1114) | Usual Care (N=1200)
Death (General disorders) | 104 (104) | 125 (125)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT02969915/Prot_SAP_000.pdf